CLINICAL TRIAL: NCT07377188
Title: Pregnancy and Inflammatory Bowel Disease
Acronym: MICI-Birth
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2019_843_0059
Record Dates: First submitted 2025-11-17; First posted 2026-01-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: IBD; Crohn's Disease; Ulcerative Colitis; Pregnancy
Keywords: IBD; Crohn's disease; Ulcerative colitis; pregnancy
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IBD and pregnancy: Population-based cohort of patients suffering from IBD and with at least one pregnancy.

SUMMARY:
Inflammatory Bowel disease, including Crohn's disease and Ulcerative Colitis, are chronic diseases.

Diagnosis is most often done in women of childbearing age. IBD can have and increase the risk of intrauterine growth retardation, preterm birth… Conversely, pregnancy can have an impact on IBD activity during pregnancy. Moreover, IBD course can be influence in post-partum. The investigators will explore IBD course on 945 patients from the EPIMAD register. The investigators will cross the data on the IBD with data on pregnancy, postpartum but also breastfeeding. The principal aim of this study is to assess the number of flares during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* women between 18 and 50 years old
* MICI diagnosed between 1988 and 2018
* included in EPIMAD registry
* living in Somme
* having had at least one pregnancy

Exclusion Criteria:

* women who has not had pregnancy
* not included in EPIMAD register

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: Patients suffering from IBD and with at least one pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 945 (Estimated)
Dates: Start 2020-09-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
number of IBD flare during pregnancy | 2 years

SECONDARY OUTCOMES:
Number of flare during post-partum period | 2 years
Number of pregnancy | 2 years
number of children | 2 years
Number of Intestinal resection | 2 years
  Intestinal resection due to mici during pregnancy and post-partum
Number of hospitalization | 2 years
  Intestinal resection and hospitalization due to mici during pregnancy and post-partum
Number of miscarriage | 2 years
Number of ectopic pregnancy | 2 years
Time before conception | 2 years
Number of women with exposition to corticosteroid | 2 years
  Exposition to corticosteroid during pregnancy and post-partum
Exposition to biotherapy | 2 years
  Exposition to biotherapy during pregnancy and post-partum
Number and indication of cesarean section | 2 years
Number of anoperineal lesions after the birth | 2 years
Wexner score for continence | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No